CLINICAL TRIAL: NCT03176615
Title: Meal-induced Thrombin Generation in Obese Women and Men Before and After Gastric Bypass - a Model of Intentional Weight Loss
Brief Title: Meal-induced Thrombin Generation Before and After Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Line Espenhain Landgrebe, Principal Investigator, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HospitalSWJ
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Morbid Obesity; Weight Loss
Keywords: Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will consume a high-fat meal and a low-fat meal served seperately in a randomized order on two seperate days (two-seven days apart)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Cross-over Group 1) (Experimental): Subjects randomly assigned to two experimental diets. This arm will receive high-fat meals first, followed by a washout period of two-seven days and then low-fat meals.
  Interventions: Dietary Supplement: Experimental diet
- Group B (Cross-over Group 2) (Experimental): Subjects randomly assigned to two experimental diets. This arm will receive low-fat meals first, followed by a washout period of two-seven days and then high-fat meals.
  Interventions: Dietary Supplement: Experimental diet

INTERVENTIONS:
Dietary Supplement: Experimental diet — The intervention will run concurrently with the gastric bypass treatment at the hospital. The first intervention is carried out before weight loss, and the intervention is repeated two times concurrently with two periods of weight loss (lifestyle and gastric bypass)

SUMMARY:
The purpose of this study is to investigate harmful effects of intentional weight loss. Intentional weight loss has been linked to increased risk of cardiovascular disease in overweight individuals, but the link between intentional weight loss and thrombotic disease is poorly understood. Postprandial coagulation activation, including thrombin generation, is a potential mechanism after high-fat meals. Thirty obese patients admitted to gastric bypass will be included in a randomized, cross-over clinical trial. All patients will consume a high-fat meal and a low-fat meal served in a randomized order on two study days (two to seven days apart). This cross-over study will be carried out before weight loss, during lifestyle-induced weight loss, and during weight loss 3-4 months after gastric bypass. Fasting and postprandial blood samples are collected on each study days, while one fecal sample is collected for each study period. The study will contribute to our understanding of mechanisms underlying harmful effects of weight loss, and future, dietary guidelines in relation to intentional weight loss programs must be modified.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for gastric bypass surgery

Exclusion Criteria:

* Use of anticoagulants, platelet inhibitors and oral contraceptives
* Known liver diseases, any malignant disorders, or known coagulation diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Postprandial peak mean of prothrombin fragment 1+2 concentrations | Measures before weight loss, change from baseline to after lifestyle-induced weight loss and 4 months post-surgery.
  Blood samples are collected after high-fat and low-fat meals on two study days.

SECONDARY OUTCOMES:
Postprandial peak mean of cardiovascular risk markers concentrations | Measures before weight loss, change from baseline to after lifestyle-induced weight loss and 4 months post-surgery.
  Blood samples are collected after high-fat and low-fat meals on two study days.
Laboratory tests of fecal samples | Measures before weight loss, change from baseline to after lifestyle-induced weight loss and 4 months post-surgery.
  Bacterial components of fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Else Bladbjerg, M.Sc. PhD, Study Chair — Unit for Thrombosis Research, Department of Regional Health Research, Hospital of South West Jutland and University of Southern Denmark
Locations (1):
- Center of Bariatric Research, Dep. of Endocrinology, Hospital of South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No